CLINICAL TRIAL: NCT01908842
Title: Induction, STabilization, Adherence, and Retention Trial (ISTART) - A Randomized, Non-inferiority, Multicenter Study to Assess Early Treatment Efficacy of OX219 Versus SUBOXONE Film and to Explore Switching Between Treatments
Brief Title: Efficacy of BNX Sublingual Tablets Versus BNX Sublingual Film for Treatment of Opioid-Dependent Adults
Acronym: ISTART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orexo AB (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OX219-006 Protocol Amendment 4
Record Dates: First submitted 2013-07-19; First posted 2013-07-26 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Opioid Dependence, on Agonist Therapy
Keywords: Opioid; Dependence; agonist; buprenorphine; naloxone; BUP/NAL
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buprenorphine; then OL BNX film, then BNX tablets (Active Comparator): Days 1-2: Generic buprenorphine sublingual tablets (blinded); Days 3 to 14: Buprenorphine/naloxone sublingual film (open-label); Days 15-21: BNX sublingual tablets (open-label); Day 22: Offered option in continuing in open-label follow-up study of BNX sublingual tablets
  Interventions: Drug: BNX sublingual tablets; Drug: BNX sublingual film; Drug: Buprenorphine
- BNX tablets, then OL BNX tablets, then BNX film (Experimental): Days 1-2: BNX sublingual tablets (blinded); Days 3 to 14: BNX sublingual tablets (open-label); Days 15-21: Buprenorphine/naloxone sublingual film (open-label); Day 22: Offered option in continuing in open-label follow-up study of BNX sublingual tablets
  Interventions: Drug: BNX sublingual tablets; Drug: BNX sublingual film

INTERVENTIONS:
Drug: BNX sublingual tablets — Buprenorphine/naloxone sublingual tablets
  Other Names: OX219; Zubsolv
Drug: BNX sublingual film — Buprenorphine/naloxone sublingual film
  Other Names: Suboxone film
Drug: Buprenorphine — Buprenorphine sublingual tablets
  Other Names: Generic buprenorphine
  Arms: Buprenorphine; then OL BNX film, then BNX tablets

SUMMARY:
The purpose of this study was to assess retention in treatment after induction with buprenorphine/naloxone (BNX) sublingual tablets compared with generic buprenorphine and after stabilization with BNX sublingual tablets compared with BNX film. Secondary objectives included assessment of treatment effects on opioid withdrawal symptoms, opioid cravings, and safety.

DETAILED DESCRIPTION:
This prospective, randomized, multicenter, parallel-group, non-inferiority study was conducted at 43 centers in the United States from August 2013 to April 2014. A non-inferior design was used because both products contain the same active components, and it was considered unethical to include a placebo arm. The study comprised an induction phase of 2 days and a stabilization phase of 20 days, with study visits scheduled on Days 1, 2, 3, 4, 8, 15, and 22. Eligible opioid-dependent patients were randomly assigned within 14 days of screening to induction with either the BNX sublingual tablets or generic buprenorphine tablets for 2 days. On Day 3, patients initially allocated to buprenorphine were switched to BNX film, whereas those allocated to BNX sublingual tablets continued on the same treatment. On Day 15, patients receiving BNX film were switched to BNX sublingual tablets, and those on BNX sublingual tablets were switched to BNX film. At the final study visit on Day 22, patients were offered the option of continuing in an open-label follow-up study of BNX sublingual tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female 18-65 years old
2. Able to read, comprehend & sign the informed consent form
3. Meet opioid dependence criteria in DSM-IV-TR the past 12 months
4. Have a buprenorphine-negative UDS &/or urine dipstick
5. Prepared to abstain from opioids other than the study drug & from other addictive drugs
6. Negative urine pregnancy test
7. Females of childbearing potential who use a reliable method of contraception. Females of non-childbearing potential; surgically sterile or post-menopausal as defined by being at least 50 years of age & having an absence of menses for at least 2 years
8. Clearance from the prescribing MD to be withdrawn from their prescribed opioids for subjects receiving opioids for pain
9. Lack of clinically significant abnormalities in health assessments performed at screening. Unclear cases should be approved by the medical monitor
10. At least mild withdrawal symptoms (COWS ≥9)

Exclusion Criteria:

1. Pregnant, lactating or planning to be pregnant during study
2. Unwilling/unable to comply with the requirements of the protocol (e.g., pending incarceration) are in a situation/condition that may interfere with participation in the study
3. Prescribed treatment with generic buprenorphine monotherapy within 90 days prior start of treatment
4. Daily dose of methadone over 30 mg during the past week or who received the last dose of methadone less than 30 hours prior to treatment
5. Participating in other clinical studies in which medications is delivered or who have used an investigational drug/device within the last 30 days
6. Allergy, sensitivity or intolerance to BUP, NAL or any related drug; history of drug hypersensitivity or intolerance which, in the opinion of the investigator, would compromise the safety of the subject/study
7. Staff, affiliated with, or family member of the staff directly involved with this study
8. Serious untreated Axis I DSM-IV-TR psychiatric comorbidity (actively suicidal or homicidal, have untreated schizophrenia)
9. Tongue/oral deformities that may affect the absorption of the drug products
10. Current/history of clinically significant medical disorder or condition which would jeopardize the safety or impact the validity of the results. Unclear cases should be discussed with & approved by the medical monitor
11. HIV-seropositive with a CD4+ count <200, active AIDS defining infection in the last 120 days
12. Have Class III/IV congestive heart failure, symptomatic myocardial ischemia or history of long QT syndrome (or an immediate family member with this condition)
13. Currently taking Class 1A antiarrhythmic medications (e.g., quinidine, procainamide, & disopyramide) or Class III antiarrhythmic medications (e.g., sotalol, amiodarone, & dofetilide)
14. Have uncontrolled hypertension, pulse oximetry ≤92%or clinically significant abnormality on 12-lead ECG, including a corrected QT (QTc) interval >450 ms
15. Severe liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Gunderson, Principal Investigator — University of Virginia, PO Box 800623, Charlottesville, VA 22911
Locations (36):
- United States (36):
  - Baldwin County, Alabama
  - Houston County, Alabama
  - Maricopa, Arizona
  - Beverly Hills, California
  - Los Angeles County, California
  - Riverside County, California
  - San Diego County, California
  - Broward County, Florida
  - Colombia County, Florida
  - Duval County, Florida
  - Greater Metro Orlando, Florida
  - Lake County, Florida
  - Miami-Dade County, Florida
  - Osceola County, Florida
  - Palm Beach County, Florida
  - DeKalb County, Georgia
  - Chicagoland, Illinois
  - Johnson County, Kansas
  - Kenton County, Kentucky
  - Caddo Parish, Louisiana
  - Baltimore County, Maryland
  - Bristol County, Massachusetts
  - Saint Louis Metro Area, Missouri
  - Camden County, New Jersey
  - Warren County, New Jersey
  - Warren County, Ohio
  - Oklahoma County, Oklahoma
  - Portland Metropolitan Area, Oregon
  - Allegheny County, Pennsylvania
  - Delaware County, Pennsylvania
  - Philadelphia County, Pennsylvania
  - Charleston County, South Carolina
  - Dallas County, Texas
  - Salt Lake County, Utah
  - Charlottesville Metropolitan Area, Virginia
  - Benton County, Washington

REFERENCES:
- [Derived] Gunderson EW, Hjelmstrom P, Sumner M; 006 Study Investigators. Effects of a higher-bioavailability buprenorphine/naloxone sublingual tablet versus buprenorphine/naloxone film for the treatment of opioid dependence during induction and stabilization: a multicenter, randomized trial. Clin Ther. 2015 Oct 1;37(10):2244-55. doi: 10.1016/j.clinthera.2015.08.025. Epub 2015 Sep 26. PMID 26412801

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 759 patients were enrolled. One patient who was randomized did not receive study drug, making the participant flow total 758.
Groups:
- BNX Tablets, Then OL BNX Tablets, Then BNX Film: Days 1-2: BNX sublingual tablets (blinded induction); Days 3 to 14: BNX sublingual tablets (open-label stabilization/maintenance); Days 15-21: Switch to BNX sublingual film (open-label stabilization/maintenance); Day 22: End of study visit
- Buprenorphine, Then OL BNX Film, Then BNX Tablets: Days 1-2: Buprenorphine (blinded induction); Days 3-14: BNX sublingual film (open-label stabilization/maintenance); Days 15-21: Switch to BNX sublingual tablets (open-label stabilization/maintenance); Day 22: End of study visit
Period: Induction
Arm/Group | BNX Tablets, Then OL BNX Tablets, Then BNX Film | Buprenorphine, Then OL BNX Film, Then BNX Tablets
Started | 383 | 375
Completed | 357 | 344
Not Completed | 26 | 31
Period: Switch to Other BNX Formulation (Day 15)
Arm/Group | BNX Tablets, Then OL BNX Tablets, Then BNX Film | Buprenorphine, Then OL BNX Film, Then BNX Tablets
Started | 357 | 344
Completed | 287 | 279
Not Completed | 70 | 65
Period: Day 22: Film (Col 1); Tablets (Col 2)
Arm/Group | BNX Tablets, Then OL BNX Tablets, Then BNX Film | Buprenorphine, Then OL BNX Film, Then BNX Tablets
Started | 287 | 279
Completed | 262 | 262
Not Completed | 25 | 17

BASELINE CHARACTERISTICS:
Groups:
- BNX Tablets, Then OL BNX Tablets, Then BNX Film: Days 1-2: BNX sublingual tablets (blinded); Days 3-14: BNX sublingual tablets (open-label); Days 15-21: Switch to BNX sublingual film (open-label); Day 22: End of study visit
- Buprenorphine, Then OL BNX Film, Then BNX Tablets: Days 1-2: Generic buprenorphine sublingual tablets (blinded); Days 3 to 14: BNX sublingual film (open-label); Days 15-21: Switch to BNX sublingual tablets (open-label); Day 22: End of study visit
- Total: Total of all reporting groups
Arm/Group | BNX Tablets, Then OL BNX Tablets, Then BNX Film | Buprenorphine, Then OL BNX Film, Then BNX Tablets | Total
Number analyzed (Participants) | 383 | 375 | 758
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (11.3) | 35.7 (11.3) | 35.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 139 | 306
  Male | 216 | 236 | 452
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 51 | 49 | 100
  White | 318 | 312 | 630
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 3 | 7 | 10
Height [Mean (Standard Deviation); unit: cm] | 171.5 (9.3) | 172.3 (9.4) | 171.9 (9.4)
Weight [Mean (Standard Deviation); unit: kg] | 77.1 (18.7) | 78.3 (18.4) | 77.7 (18.6)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 26.2 (5.9) | 26.3 (5.7) | 26.3 (5.8)
Duration of opioid use [Mean (Standard Deviation); unit: years] | 10.7 (9.6) | 10.5 (9.0) | 10.6 (9.3)

OUTCOME MEASURES:

1. Secondary Outcome: Clinical Opiate Withdrawal Scale (COWS) Scores: Induction
Description: Absolute ± mean standard deviation values for COWS total scores at baseline; 0.5 h, 1.5 h, 3 h, and 6 h post dose on Day 1, and Day 2; COWS scores range from 0-48, with a lower score being more favorable
Time Frame: Days 1 and 2
Population: Full Analysis Population - number of enrolled patients at the beginning of the measurement period
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- BNX Tablets, Then OL BNX Tablets, Then BNX Film: Days 1-2: BNX sublingual tablets (blinded induction); Days 3-14: BNX sublingual tablets (open-label stabilization/maintenance); Days 15-21: Switch to BNX sublingual film (open-label stabilization/maintenance); Day 22: End of study visit
- Buprenorphine, Then OL BNX Film, Then BNX Tablets: Days 1-2: Buprenorphine sublingual tablets (blinded induction); Days 3-14: BNX sublingual film (open-label stabilization/maintenance); Days 15-21: Switch to BNX sublingual tablets (open-label stabilization/maintenance); Day 22: End of study visit
Arm/Group | BNX Tablets, Then OL BNX Tablets, Then BNX Film | Buprenorphine, Then OL BNX Film, Then BNX Tablets
Number analyzed (Participants) | 380 | 373
units on a scale
  Baseline | 15.0 (4.2) | 14.9 (4.3)
  Day 1 0.5 h post dose | 10.5 (4.6) | 10.3 (4.7)
  Day 1 1.5 h post dose | 8.8 (4.6) | 8.3 (4.5)
  Day 1 3 h post dose | 6.6 (5.1) | 6.1 (5.1)
  Day 1 6 h post dose | 5.3 (4.1) | 5.4 (4.6)
  Day 2 | 8.0 (4.9) | 7.6 (5.2)

2. Secondary Outcome: COWS Total Scores: Stabilization/Maintenance
Description: Absolute ± mean standard deviation values for COWS total scores at Days 3, 4, 8, 15, and 22; COWS scores range from 0-48, with a lower score being more favorable
Time Frame: Days 3 through 22
Population: Full analysis population - - number of enrolled patients at the beginning of the measurement period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BNX Tablets, Then OL BNX Tablets, Then BNX Film | Buprenorphine, Then OL BNX Film, Then BNX Tablets
Number analyzed (Participants) | 355 | 344
units on a scale
  Day 3 | 6.0 (4.2) | 5.9 (4.4)
  Day 4 | 5.2 (4.0) | 5.1 (4.3)
  Day 8 | 4.8 (3.9) | 4.6 (3.9)
  Day 15 | 4.1 (3.5) | 3.7 (3.4)
  Day 22: Film (col 1); Tablets (col 2) | 3.4 (3.3) | 3.3 (3.4)

3. Secondary Outcome: Subjective Opiate Withdrawal Scale (SOWS) Scores: Induction
Description: Absolute ± mean standard deviation values for SOWS total scores at baseline, 0.5 h, 1.5 h, 3 h, and 6 h post dose on Day 1, and Day 2; SOWS score ranges from 0-64, with a lower score being more favorable
Time Frame: Days 1 and 2
Population: Full analysis population - number of enrolled patients at the beginning of the measurement period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BNX Tablets, Then OL BNX Tablets, Then BNX Film | Buprenorphine, Then OL BNX Film, Then BNX Tablets
Number analyzed (Participants) | 376 | 367
units on a scale
  Baseline | 31.7 (13.5) | 33.0 (13.2)
  Day 1 0.5 h post dose | 22.7 (13.9) | 23.0 (13.6)
  Day 1 1.5 h post dose | 19.1 (13.5) | 17.8 (13.0)
  Day 1 3 h post dose | 13.6 (12.7) | 13.0 (12.5)
  Day 1 6 h post dose | 10.7 (10.2) | 11.1 (11.8)
  Day 2 | 16.7 (12.3) | 16.4 (13.4)

4. Primary Outcome: Primary Endpoints of Retention in Treatment at Days 3 and 15
Description: Retention rates (number of patients retained) for the primary efficacy endpoints of retention in treatment at Days 3 and 15, which was defined as the number of patients who received treatment on Days 3 and 15.
Time Frame: Day 3 and Day 15
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | BNX Tablets, Then OL BNX Tablets, Then BNX Film | Buprenorphine, Then OL BNX Film, Then BNX Tablets
Number analyzed (Participants) | 329 | 326
participants
  Retention at Day 3 | 309 | 302
  Retention at Day 15 | 273 | 269

5. Secondary Outcome: SOWS Total Scores: Stabilization/Maintenance
Description: Absolute ± mean standard deviation values for SOWS total scores on Days 2, 3, 4, 8, 15, and 22; SOWS scores ranged from 0-64, with a lower score being more favorable
Time Frame: Days 3 through 22
Population: Full Analysis Population - number of enrolled patients at the beginning of the measurement period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BNX Tablets, Then OL BNX Tablets, Then BNX Film | Buprenorphine, Then OL BNX Film, Then BNX Tablets
Number analyzed (Participants) | 355 | 342
units on a scale
  Day 3 | 11.9 (10.4) | 12.6 (11.2)
  Day 4 | 10.1 (9.2) | 10.2 (10.3)
  Day 8 | 9.0 (9.2) | 8.8 (9.6)
  Day 15 | 7.2 (7.7) | 6.7 (8.1)
  Day 22: Film (col 1); Tablets (col 2) | 6.8 (7.9) | 7.3 (9.2)

6. Secondary Outcome: Visual Analog Scale (VAS) Cravings: Induction
Description: Absolute mean ± standard deviation values for VAS cravings at baseline, 0.5 h, 1.5 h, 3 h, and 6 post dose on Day 1, and Day 2; the VAS craving scores range from 0 ("no cravings") to 100 ("most intense craving I have ever had")
Time Frame: Days 1 and 2
Population: Full Analysis Population - number of enrolled patients at the beginning of the measurement period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BNX Tablets, Then OL BNX Tablets, Then BNX Film | Buprenorphine, Then OL BNX Film, Then BNX Tablets
Number analyzed (Participants) | 380 | 373
units on a scale
  Baseline | 69.2 (23.5) | 71.9 (22.0)
  Day 1 0.5 h post dose | 56.8 (26.5) | 58.2 (26.4)
  Day 1 1.5 h post dose | 49.2 (28.9) | 48.8 (27.9)
  Day 1 3 h post dose | 36.0 (28.2) | 34.9 (27.8)
  Day 1 6 h post dose | 30.2 (26.2) | 29.6 (26.9)
  Day 2 | 45.3 (28.7) | 44.9 (28.4)

7. Secondary Outcome: VAS Craving Scores: Stabilization/Maintenance
Description: Absolute mean ± standard deviation values for VAS cravings scores on Days 3, 4, 8, 15, and 22; the VAS craving scores range from 0 ("no cravings") to 100 ("most intense craving I have ever had")
Time Frame: Days 3 through 22
Population: Full analysis population - number of enrolled patients at the beginning of the measurement period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BNX Tablets, Then OL BNX Tablets, Then BNX Film | Buprenorphine, Then OL BNX Film, Then BNX Tablets
Number analyzed (Participants) | 356 | 344
units on a scale
  Day 3 | 33.7 (27.0) | 34.5 (28.2)
  Day 4 | 29.1 (26.2) | 28.5 (26.4)
  Day 8 | 26.2 (26.5) | 23.7 (24.7)
  Day 15 | 21.6 (23.9) | 19.1 (23.4)
  Day 22: Film (col 1); Tablets (col 2) | 20.2 (22.9) | 20.9 (23.8)

ADVERSE EVENTS:
Time Frame: Monitoring for adverse events was conducted from baseline through Day 22.
Arm/Group | BNX Tablets, Then OL BNX Tablets, Then BNX Film | Buprenorphine, Then OL BNX Film, Then BNX Tablets
Serious Adverse Events (participants affected / at risk) | 3/383 | 1/375
Other Adverse Events (participants affected / at risk) | 61/383 | 55/375
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNX Tablets, Then OL BNX Tablets, Then BNX Film (N=383) | Buprenorphine, Then OL BNX Film, Then BNX Tablets (N=375)
Worsening of pre-existing condition (foreign body in neck) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Serious adverse event reported during blinded induction phase.
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Serious adverse event reported during open-label maintenance phase.
Elevated Transaminases (Hepatobiliary disorders) | 1 (1) | 0 (0) — Serious adverse event reported during open-label maintenance phase.
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) — Serious adverse event reported during blinded induction phase.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNX Tablets, Then OL BNX Tablets, Then BNX Film (N=383) | Buprenorphine, Then OL BNX Film, Then BNX Tablets (N=375)
Headache (Nervous system disorders) | 20 (20) | 19 (19) — Adverse events reported during the blinded induction phase.
Vomiting (Gastrointestinal disorders) | 12 (12) | 11 (11) — Adverse events reported during the blinded induction phase.
Nausea (Gastrointestinal disorders) | 8 (8) | 15 (15) — Adverse events reported during the blinded induction phase.
Dry mouth (Gastrointestinal disorders) | 8 (8) | 2 (2) — Adverse events reported during the blinded induction phase.
Insomnia (Psychiatric disorders) | 5 (5) | 4 (4) — Adverse events reported during the blinded induction phase.
Somnolence (Nervous system disorders) | 6 (6) | 2 (2) — Adverse events reported during the blinded induction phase.
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3) — Adverse events reported during the blinded induction phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No